CLINICAL TRIAL: NCT01818102
Title: CT Window Setting to Select Double-lumen Tube Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JHBahk_DLT_CT window
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Bronchial Cuff Volume at Air-tight Seal; Intracuff Cuff Pressure at Air-tighe Seal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Width 1000 HU/Level -450 HU (Experimental)
  Interventions: Device: Width 1000 HU/Level -450 HU
- Width 400 HU/Level 25 HU (Active Comparator)
  Interventions: Device: Width 400 HU/Level 25 HU

INTERVENTIONS:
Device: Width 1000 HU/Level -450 HU — Double-lumen tube size is selected according to the internal diameter of the left mainstem bronchus measured in the chest computed tomography with width 1000 HU and level -450 HU.
  Arms: Width 1000 HU/Level -450 HU
Device: Width 400 HU/Level 25 HU — Double-lumen tube size is selected according to the internal diameter of the left mainstem bronchus measured in the chest computed tomography with width 400 HU and level 25 HU.
  Arms: Width 400 HU/Level 25 HU

SUMMARY:
The purpose of this study is to investigate the appropriate window setting of chest computed tomography to select a correct size of double-lumen endobronchial tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that require the placement of left-sided double-lumen tubes

Exclusion Criteria:

* Abnoraml anatomy of tracheobronchail tree
* Intraluminal lesion in the left mainstem bronchus
* Anticipated difficult intubation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Air-leak at deflation of bronchial cuff | An expected average of 10 min after double lumen tube intubation
Air-tight seal below resting volume of bronchial cuff | An expected average of 10 min after double lumen tube intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea